CLINICAL TRIAL: NCT04181099
Title: Influence of Different Zirconia Surface Treatments on Biofilm Formation
Acronym: Biofilm2020
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Basel (Other)
Responsible Party: Principal Investigator, Nadja Rohr, Principal Investigator, University of Basel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019-01918
Record Dates: First submitted 2019-11-26; First posted 2019-11-29 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Surface Finish
Keywords: dental implant; zirconia; biofilm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zirconia structure (Other): The participants will carry an orthodontic device containing 4 discs of differently structured zirconia and titanium to test the biofilm formation in order to determine the ideal structure for the neck area of zirconia dental implants.
  Interventions: Other: Implant neck surface

INTERVENTIONS:
Other: Implant neck surface — The biofilm formation is tested on discs manufactured of zirconia with different surfaces in vivo using orthodontic devices that the participants carry over 24h

SUMMARY:
The aim is to test the influence of surface finish on biofilm formation on the transmucosal part of zirconia implants in an in vivo study. Sixteen test person will therefore receive an orthodontic apparatus containing the specimens with the respective surfaces and carry them for 2x 24h. The primary outcome is the spectormetrical quantification (OD value) of biofilm on the specimens that have been carried by the test person over 24h. Biofilm will be analysed using scanning electron microscopy.

ELIGIBILITY:
Inclusion Criteria:

* No systematic antibiotic therapy during the last 3 months
* Good oral health and compliance (PI and BI <20%)
* No sign of parodontal disease or other inflammatory changes in the mouth
* Non-smoker

Exclusion Criteria:

* Disease that requires antibiotic therapy
* Pressure marks due to the orthodontic apparatus that can not be eliminated
* Other unexpected complications that could be related to the orthodontic apparatus

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Safranin Staining | 3 months
  The biofilm on the discs is quantified using safranin staining and evaluated with the measurement of optical density using a photospectrometer

SECONDARY OUTCOMES:
SEM | 3 months
  The morphology of the biofilm is analyzed using scanning electron microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Jens Fischer, Prof, Study Director — University Center for Dental Medicine Basel
Locations (1):
- University Center for Dental Medicine Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No